CLINICAL TRIAL: NCT03457857
Title: A Single Center, Five Week, Evaluator Blinded, Clinical Trial Evaluating Two Cleansing and/or Moisturizing Regimens on the Skin of Healthy Infants Using Clinical, Instrumental, D-Squame Tape, Microbiome and Parental Assessments
Brief Title: Evaluation of Two Regimens, With Healthy Male and Female Babies, Ages 3-6 Months Old, Using Various Assessments.
Acronym: Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CO-170929100633-SBCT
Record Dates: First submitted 2018-02-01; First posted 2018-03-08 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Microbiome
Keywords: Microbiome; Microbiota

STUDY DESIGN:
Intervention Model Description: The duration of this trial will be approximately 5 weeks and will consist of a screening visit followed by an approximately 1-week (7-day) washout period; a 4-week (28 day) treatment period with visits conducted at baseline (Day 0, ± 2 days), week 2 (Day 14, ± 2 days), and week 4 (Day 28, ± 2 days); and a regression period with a visit 3-5 days after the week 4 visit.
  During the one week washout period, subjects will use a commercial available Baby Wash at least 3x per week.
  For the next 4 weeks, subjects will be randomly assigned to use one of two IP regiments. Subjects in Group 1 will use the Baby Wash & Shampoo at least 3x per week, but no more than once daily. Subjects in Group 2 will use the Baby Wash & Shampoo at least 3x per week, but no more than once daily, plus the Baby Lotion at least once daily. The lotion should be applied after bathing (as applicable).
  At Visit 4, subjects will begin a 3-5 day regression period.
Who Masked: Investigator
Masking Description: This study will be evaluator-blinded, so the PI/expert graders will not know which group (Group 1 or Group 2) each subject is in. Personnel dispensing the IPs or supervising IP use will not participate in the evaluation of subjects in order to minimize potential bias. IPs will be kept separate from the site personnel involved in assessing or evaluating the subjects, and subjects will be instructed not to discuss their assigned IPs with the PI/expert graders or other subjects.
  To keep the evaluator blinded, the study staff will keep the grading forms separate from the bulk of the source documents so the evaluator will not have access to the sheets that indicate randomization and the study staff will instruct the subjects/LAR to not say anything about what product they are using.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Cleanser (Other): Regimen with Baby Cleanser Only
  Interventions: Other: Cleanser
- Group 2 - Cleanser and Lotion (Other): Regimen containing Baby Cleanser/Shampoo and Baby Lotion
  Interventions: Other: Cleanser and Lotion

INTERVENTIONS:
Other: Cleanser — Cosmetic Baby Cleanser/Shampoo
  Arms: Group 1 - Cleanser
Other: Cleanser and Lotion — Cosmetic Baby Cleanser/Shampoo and Baby Lotion
  Arms: Group 2 - Cleanser and Lotion

SUMMARY:
This study is to assess the impact of two skincare regimens on the cutaneous microbiome and skin physiology of healthy male and female infants, ages 3-6 months using clinical, instrumental, D-Squame tape, microbiome and parental assessments over a five-week period.

DETAILED DESCRIPTION:
Skin cleansing has been demonstrated as a simple strategy to help keep skin healthy. There are many types of cleansing and moisturizing routines that have been shown to have different effects on the skin barrier such as reducing sebum and exogenous contaminants, controlling odors, and affecting the skin microbiome.1 A previous study in an adult population showed that use of a mild surfactant cleanser had less of an impact on the skin barrier than a liquid castile soap (data on file ).2 Because infant skin differs from an adult's in structure, function, and composition3, cleanser and/or lotion regimens may impact the skin barrier of infants differently.

There is very little information in the literature on how the use of product regimens impacts the cutaneous microbiome and skin physiology of adults1 and even less about how it impacts the skin of children.

This study will explore the impact that the use of two regimens - one cleansing and the other cleansing and moisturizing - has on the holistic skin barrier of infants ages 3-6 months.

The IPs are a baby wash and a baby lotion, which are both cosmetic body products. The auxiliary product is a commercially available, cosmetic baby body wash.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* 3 - 6 months old (up to but not including 7 months, 0 days)
* Generally in good health based on medical history reported by the subject's parent/LAR.
* Parent/LAR Is 18 years of age or older and willing/able to present proof of guardianship for the infant subject (i.e., birth certificate, hospital records, adoption record, insurance card, other ID along with valid ID of parent/LAR).
* Parent/LAR has signed the ICD including Health Insurance Portability and Accountability Act (HIPAA) disclosure in English, for the infant to participate in the study.
* Parent/LAR agrees not to introduce any new products or fragrances on his/her person, on his/her infant (e.g. cleansers, lotions, perfumes, etc.), or in the household environment that the infant may come in contact with (e.g. room fresheners, cleansing agents, etc.) for the duration of the study other than the product provided.
* Parent/LAR agrees to limit subject's sun exposure and to use appropriate sun protection including clothing, hats and shade as appropriate. Subject's own sunscreen may be used at the parent's/LAR's discretion on exposed areas, but use should be documented. Parent/LAR should make every effort to limit the subject's sun exposure for the duration of the study.
* Parent/LAR is willing and able to participate in and comply with the study requirements including using the investigational study materials as directed on his/her infant throughout the study period.
* Parent/LAR agrees not to use the provided products on self or any family member other than the infant subject.
* Parent/LAR agrees to not allow their infant to participate in another clinical study or product use study during the study duration.
* Parent/LAR agrees to the possible subsequent use of the data in medical or scientific journals and medical or scientific presentation materials and advertising materials. All subject identities will remain confidential.

Exclusion Criteria

* Has known allergies, adverse reactions, or unusual hypersensitivity to common topical skincare products or their components, fragrances, skin care toiletry products or adhesive tapes.
* Presents with a skin condition that may influence the outcome of the study (specifically psoriasis, eczema, atopic dermatitis, cutaneous xerosis, erythema, active skin cancer, sensitive skin, moderate to severe looking diaper rash).
* Actively taking any medications, particularly antibiotics either oral or topical, as they may interfere with the study. Any condition requiring use of a topical or oral OTC or prescription medication, which in the Study Physician's judgement makes the subject ineligible or places the subject at risk (e.g. antibiotics such as Amoxicillin, Zithromax, Cefphalexin or any other medications that may cause gastrointestinal distress/diarrhea that will affect skin condition/cause irritation/rash of genital/buttocks area).
* Infant may not swim, or use hot tubs or pools for the duration of the study.
* Has Type 1 or Type 2 diabetes or is taking insulin or another anti-diabetic medication as reported by the parent/LAR.
* Has taken medications that would mask an AE or influence the study results, including:

  * Immunosuppressive drugs and steroidal and/or non-steroidal anti-inflammatory drugs within 3 months before Visit 1 and during the study.
  * Antihistamines within 1 month before Visit 1 and during the study.
  * Receiving systemic or topical medications, which may interfere with study evaluations.
  * Has a history of or a concurrent health condition/situation, which, in the opinion of the PI or Study Physician, may put the individual at significant risk, confound the study results, or interfere significantly with the individual's participation in the study.
* Is simultaneously participating in any other type of clinical study or product use study
* Has had a recent change in dietary intake within 1 week (7 days) prior to study start.
* Has a known condition of asthma or any related breathing problem and/or for whom there is a family history of asthma.
* Has an active localized or general infections including upper respiratory infections (ear, nose, throat, fever, cough, etc.).
* Has excessive scars, which could interfere with expert grader evaluations.
* Is viewed by the PI or Study Physician as not being able to complete the study.
* Parent/LAR is pregnant and/or planning to become pregnant during the study or within the next 3 months.

Ages: 3 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
Change in Skin hydration values | Change in skin hydration values from Baseline (Day 0) to Day 28.
  Skin hydration as assessed by mean Corneometer measurements on the dorsal forearm. Group 2 with baby lotion will also be assessed by dry down of lotion at Baseline (Day 0)
Change in Skin pH values | Change in skin pH values from Baseline (Day 0) to Day 28.
  Skin pH as assessed by mean skin pH on the dorsal forearm at all time points. Group 2 with baby lotion only will be assessed after dry down of the lotion at Baseline (Day 0)
Change in Skin hydration values | Change in skin hydration values from Baseline (Day 0) to Day 14.
  Skin hydration as assessed by mean Corneometer measurements on the dorsal forearm. Group 2 with baby lotion will also be assessed by dry down of lotion at Baseline (Day 0)
Change in Skin hydration values | Change in skin hydration values from post-baseline (regression) minus Baseline (Day 0) to Day 28.
  Skin hydration as assessed by mean Corneometer measurements on the dorsal forearm. Group 2 with baby lotion will also be assessed by dry down of lotion at Baseline (Day 0)
Change in Skin hydration values | Change in skin hydration values from post-baseline (regression) minus Baseline (Day 0) to Day 14.
  Skin hydration as assessed by mean Corneometer measurements on the dorsal forearm. Group 2 with baby lotion will also be assessed by dry down of lotion at Baseline (Day 0)
Change in Skin pH values | Change in skin pH values from Baseline (Day 0) to Day 14.
  Skin pH as assessed by mean skin pH on the dorsal forearm at all time points. Group 2 with baby lotion only will be assessed after dry down of the lotion at Baseline (Day 0)
Change in Skin pH values | Change in skin pH values from post-baseline (regression) minus Baseline (Day 0) to Day 28.
  Skin pH as assessed by mean skin pH on the dorsal forearm at all time points. Group 2 with baby lotion only will be assessed after dry down of the lotion at Baseline (Day 0)
Change in Skin pH values | Change in skin pH values from post-baseline (regression) minus Baseline (Day 0) to Day 14.
  Skin pH as assessed by mean skin pH on the dorsal forearm at all time points. Group 2 with baby lotion only will be assessed after dry down of the lotion at Baseline (Day 0)

SECONDARY OUTCOMES:
Change in Overall Skin Appearance (Evaluated by PI) | Change in Overall Skin Appearance from Baseline (Day 0) to Day 28
  Overall Skin Appearance on a 10 Point Scale from Poor (Score =1) to Excellent (Score =10)
Change in Overall Skin Appearance (Evaluated by parent/LAR) | Change in Overall Skin Appearance from Baseline (Day 0) to Day 28.
  Overall Skin Appearance will be evaluated by the parent/LAR on a 10-point Scale ranging from Poor (Score =1) to Excellent (Score =10)
D-Squame Tapes | Baseline (Day 0) and Day 28
  D-Squame Tape samples will be taken on the dorsal forearm, which safely removes stratum corneum components, visibility of adhering corneocytes and a metabolomics method.
Microbial Community Richness | Baseline (Day 0), Day 14, Day 28 and 3-5 days Regression
  Microbial Community Richness on the forehead, dorsal forearm and buttock based on the total number of different bacterial taxa detected in the sample.
Microbial Community Diversity | Baseline (Day 0), Day 14, Day 28 and 3-5 days Regression
  Microbial Community Diversity on the forehead, dorsal forearm and buttock based on the Shannon Index.
Microbial Community Evenness | Baseline (Day 0), Day 14, Day 28 and 3-5 days regression
  Microbial Community Evenness on the forehead, dorsal forearm and buttock based on Pielou's evenness index.
Change in Clinical Assessment Evaluation for Dryness (Evaluated by PI) | Change in Dryness Scores from Baseline (Day 0) to Day 28.
  Clinical Assessments for Dryness will be evaluated on a 4-point Scale from 0 = None, 1 = Mild, 2 = Moderate and 3= Severe globally by the PI
Change in Overall Skin Appearance (Evaluated by PI) | Change in Overall Skin Appearance from Baseline (Day 0) to Day 14
  Overall Skin Appearance on a 10 Point Scale from Poor (Score =1) to Excellent (Score =10)
Change in Overall Skin Appearance (Evaluated by PI) | Change in Overall Skin Appearance from Baseline (Day 0) to Regression (3-5 Days)
  Overall Skin Appearance on a 10 Point Scale from Poor (Score =1) to Excellent (Score =10)
Change in Overall Skin Appearance (Evaluated by parent/LAR) | Change in Overall Skin Appearance from Baseline (Day 0) to Regression (3-5 Days)
  Overall Skin Appearance will be evaluated by the parent/LAR on a 10-point Scale ranging from Poor (Score =1) to Excellent (Score =10)
Change in Overall Skin Appearance (Evaluated by parent/LAR) | Change in Overall Skin Appearance from Baseline (Day 0) to Day 14.
  Overall Skin Appearance will be evaluated by the parent/LAR on a 10-point Scale ranging from Poor (Score =1) to Excellent (Score =10)
Change in Clinical Assessment Evaluation for Dryness (Evaluated by PI) | Change in Dryness Scores from Baseline (Day 0) to Day 14.
  Clinical Assessments for Dryness will be evaluated on a 4-point Scale from 0 = None, 1 = Mild, 2 = Moderate and 3= Severe globally by the PI
Change in Clinical Assessment Evaluation for Dryness (Evaluated by PI) | Change in Dryness Scores from Baseline (Day 0) to Regression (3-5 Days).
  Clinical Assessments for Dryness will be evaluated on a 4-point Scale from 0 = None, 1 = Mild, 2 = Moderate and 3= Severe globally by the PI
Change in Clinical Assessment Evaluation for Redness/Erythema (Evaluated by PI) | Change in Redness/Erythema Scores from Baseline (Day 0) to Day 28.
  Clinical Assessments for Redness/Erythema will be evaluated on a 4-point Scale from 0 = None, 1 = Mild, 2 = Moderate and 3= Severe globally by the PI
Change in Clinical Assessment Evaluation for Redness/Erythema (Evaluated by PI) | Change in Redness/Erythema Scores from Baseline (Day 0) to Day 14.
  Clinical Assessments for Redness/Erythema will be evaluated on a 4-point Scale from 0 = None, 1 = Mild, 2 = Moderate and 3= Severe globally by the PI
Change in Clinical Assessment Evaluation for Redness/Erythema (Evaluated by PI) | Change in Redness/Erythema Scores from Baseline (Day 0) to Regression (3-5 Days).
  Clinical Assessments for Redness/Erythema will be evaluated on a 4-point Scale from 0 = None, 1 = Mild, 2 = Moderate and 3= Severe globally by the PI
Change in Clinical Assessment Evaluation for Rash/Irritation (Evaluated by PI) | Change in Rash/Irritation Scores from Baseline (Day 0) to Day 28.
  Clinical Assessments for Rash/Irritation will be evaluated on a 4-point Scale from 0 = None, 1 = Mild, 2 = Moderate and 3= Severe globally by the PI
Change in Clinical Assessment Evaluation for Rash/Irritation (Evaluated by PI) | Change in Rash/Irritation Scores from Baseline (Day 0) to Day 14.
  Clinical Assessments for Rash/Irritation will be evaluated on a 4-point Scale from 0 = None, 1 = Mild, 2 = Moderate and 3= Severe globally by the PI
Change in Clinical Assessment Evaluation for Rash/Irritation (Evaluated by PI) | Change in Rash/Irritation Scores from Baseline (Day 0) to Regression (3-5 Days)
  Clinical Assessments for Rash/Irritation will be evaluated on a 4-point Scale from 0 = None, 1 = Mild, 2 = Moderate and 3= Severe globally by the PI
Change in Clinical Assessment Evaluation for Tactile Roughness (Evaluated by PI) | Change in Tactile Roughness Scores from Baseline (Day 0) to Day 28.
  Clinical Assessments for Tactile Roughness will be evaluated on a 4-point Scale from 0 = None, 1 = Mild, 2 = Moderate and 3= Severe globally by the PI
Change in Clinical Assessment Evaluation for Tactile Roughness (Evaluated by PI) | Change in Tactile Roughness Scores from Baseline (Day 0) to Day 14.
  Clinical Assessments for Tactile Roughness will be evaluated on a 4-point Scale from 0 = None, 1 = Mild, 2 = Moderate and 3= Severe globally by the PI
Change in Clinical Assessment Evaluation for Tactile Roughness (Evaluated by PI) | Change in Tactile Roughness Scores from Baseline (Day 0) to Regression (3-5 Days).
  Clinical Assessments for Tactile Roughness will be evaluated on a 4-point Scale from 0 = None, 1 = Mild, 2 = Moderate and 3= Severe globally by the PI
Change in Skin Irritation (Evaluated by PI) | Change in Skin Irritation from Baseline (Day 0) to Day 28
  Skin Irritation will be evaluated by the PI on a 10 Point Scale from Very Irritated (Score =1) to Not Irritated (Score =10)
Change in Skin Irritation (Evaluated by PI) | Change in Skin Irritation from Baseline (Day 0) to Day 14
  Skin Irritation will be evaluated by the PI on a 10 Point Scale from Very Irritated (Score =1) to Not Irritated (Score =10)
Change in Skin Irritation (Evaluated by PI) | Change in Skin Irritation from Baseline (Day 0) to Regression (3-5 Days)
  Skin Irritation will be evaluated by the PI on a 10 Point Scale from Very Irritated (Score =1) to Not Irritated (Score =10)
Change in Skin Irritation (Evaluated by parent/LAR) | Change in Skin Irritation from Baseline (Day 0) to Day 28
  Skin Irritation will be evaluated by the parent/LAR on a 10 Point Scale from Very Irritated (Score =1) to Not Irritated (Score =10)
Change in Skin Irritation (Evaluated by parent/LAR) | Change in Skin Irritation from Baseline (Day 0) to Day 14
  Skin Irritation will be evaluated by the parent/LAR on a 10 Point Scale from Very Irritated (Score =1) to Not Irritated (Score =10)
Change in Skin Irritation (Evaluated by parent/LAR) | Change in Skin Irritation from Baseline (Day 0) to Regression (3-5 Days)
  Skin Irritation will be evaluated by the parent/LAR on a 10 Point Scale from Very Irritated (Score =1) to Not Irritated (Score =10)
Change in Skin Dryness (Evaluated by PI) | Change in Skin Dryness from Baseline (Day 0) to Day 28
  Skin Dryness will be evaluated by the PI on a 10 Point Scale from Very Dry (Score =1) to No Visible Dryness (Score =10)
Change in Skin Dryness (Evaluated by PI) | Change in Skin Dryness from Baseline (Day 0) to Day 14.
  Skin Dryness will be evaluated by the PI on a 10 Point Scale from Very Dry (Score =1) to No Visible Dryness (Score =10)
Change in Skin Dryness (Evaluated by PI) | Change in Skin Dryness from Baseline (Day 0) to Regression (3-5 Days)
  Skin Dryness will be evaluated by the PI on a 10 Point Scale from Very Dry (Score =1) to No Visible Dryness (Score =10)
Change in Skin Dryness (Evaluated by parent/LAR) | Change in Skin Dryness from Baseline (Day 0) to Day 28
  Skin Dryness will be evaluated by the parent/LAR on a 10 Point Scale from Very Dry (Score =1) to No Visible Dryness (Score =10)
Change in Skin Dryness (Evaluated by parent/LAR) | Change in Skin Dryness from Baseline (Day 0) to Day 14.
  Skin Dryness will be evaluated by the parent/LAR on a 10 Point Scale from Very Dry (Score =1) to No Visible Dryness (Score =10)
Change in Skin Dryness (Evaluated by parent/LAR) | Change in Skin Dryness from Baseline (Day 0) to Regression (3-5 Days)
  Skin Dryness will be evaluated by the parent/LAR on a 10 Point Scale from Very Dry (Score =1) to No Visible Dryness (Score =10)
Change in Skin Softness (Evaluated by PI) | Change in Skin Softness from Baseline (Day 0) to Day 28
  Skin Softness will be evaluated by the PI on a 10 Point Scale from Not Soft (Score =1) to Very Soft (Score =10)
Change in Skin Softness (Evaluated by PI) | Change in Skin Softness from Baseline (Day 0) to Day 14
  Skin Softness will be evaluated by the PI on a 10 Point Scale from Not Soft (Score =1) to Very Soft (Score =10)
Change in Skin Softness (Evaluated by PI) | Change in Skin Softness from Baseline (Day 0) to Regression (3-5 Days)
  Skin Softness will be evaluated by the PI on a 10 Point Scale from Not Soft (Score =1) to Very Soft (Score =10)
Change in Skin Softness (Evaluated by parent/LAR) | Change in Skin Softness from Baseline (Day 0) to Day 28
  Skin Softness will be evaluated by the parent/LAR on a 10 Point Scale from Not Soft (Score =1) to Very Soft (Score =10)
Change in Skin Softness (Evaluated by parent/LAR) | Change in Skin Softness from Baseline (Day 0) to Day 14.
  Skin Softness will be evaluated by the parent/LAR on a 10 Point Scale from Not Soft (Score =1) to Very Soft (Score =10)
Change in Skin Softness (Evaluated by parent/LAR) | Change in Skin Softness from Baseline (Day 0) to Regression (3-5 Days)
  Skin Softness will be evaluated by the parent/LAR on a 10 Point Scale from Not Soft (Score =1) to Very Soft (Score =10)
Change in Skin Roughness (Evaluated by PI) | Change in Skin Roughness from Baseline (Day 0) to Day 28
  Skin Roughness will be evaluated by the PI on a 10 Point Scale from Very Rough (Score =1) to Very Smooth (Score =10)
Change in Skin Roughness (Evaluated by PI) | Change in Skin Roughness from Baseline (Day 0) to Day 14.
  Skin Roughness will be evaluated by the PI on a 10 Point Scale from Very Rough (Score =1) to Very Smooth (Score =10)
Change in Skin Roughness (Evaluated by PI) | Change in Skin Roughness from Baseline (Day 0) to Regression (3-5 Days)
  Skin Roughness will be evaluated by the PI on a 10 Point Scale from Very Rough (Score =1) to Very Smooth (Score =10)
Change in Skin Roughness (Evaluated by parent/LAR) | Change in Skin Roughness from Baseline (Day 0) to Day 28
  Skin Roughness will be evaluated by the parent/LAR on a 10 Point Scale from Very Rough (Score =1) to Very Smooth (Score =10)
Change in Skin Roughness (Evaluated by parent/LAR) | Change in Skin Roughness from Baseline (Day 0) to Day 14
  Skin Roughness will be evaluated by the parent/LAR on a 10 Point Scale from Very Rough (Score =1) to Very Smooth (Score =10)
Change in Skin Roughness (Evaluated by parent/LAR) | Change in Skin Roughness from Baseline (Day 0) to Regression (3-5 Days)
  Skin Roughness will be evaluated by the parent/LAR on a 10 Point Scale from Very Rough (Score =1) to Very Smooth (Score =10)

OTHER OUTCOMES:
Number of participants who provide information about their families at Day 31 - Day 33 (Regression) | Questionnaire Data from Day 31 to Day 33
  Parent/LAR will complete a questionnaire about Breastfeeding, Delivery, Touch and Environment. There are no baseline measures for comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Jumbelic, BS, Principal Investigator — SourceOne Technical Solution
Locations (1):
- Johnson & Johnson Consumer Experience Center, Skillman, New Jersey, United States

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CO-170929100633-SBCT&attachmentIdentifier=1f64b222-2756-46c9-9beb-36c885fdc2f3&fileName=Summary_CSR_for_Rembrandt_Microbiome_06_Aug_2019_Redacted.pdf&versionIdentifier=